CLINICAL TRIAL: NCT00064012
Title: A Randomized, Multicenter, Open-Label, Phase II Study Of VELCADE Alone Or VELCADE Plus Docetaxel In Previously Treated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Bortezomib With or Without Docetaxel in Treating Patients With Relapsed or Refractory Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000305974; P30CA016042 (NIH); WCCC-M34102-048; UCLA-0301037; MILLENNIUM-M34102-048
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2013-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib; Docetaxel

ARMS (2):
- Velcade Alone (Active Comparator): Velcade
  Interventions: Drug: bortezomib
- Velcade plus Docetaxel (Experimental): Velcade plus Docetaxel
  Interventions: Drug: bortezomib; Drug: docetaxel

INTERVENTIONS:
Drug: bortezomib
Drug: docetaxel
  Arms: Velcade plus Docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as docetaxel use different ways to stop tumor cells from dividing so they stop growing or die. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. It is not yet known whether bortezomib is more effective with or without docetaxel in treating patients with advanced non-small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of bortezomib with or without docetaxel in treating patients who have relapsed or refractory stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the tumor response rates (complete and partial response) in patients with relapsed or refractory advanced non-small cell lung cancer treated with bortezomib with vs without docetaxel.

Secondary

* Compare time to progression in patients treated with these regimens.
* Compare the overall and 1-year survival of patients treated with these regimens.
* Compare the safety and tolerability of these regimens in these patients.
* Compare the pharmacokinetics and pharmacodynamics of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1 and bortezomib IV as in arm I.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses beyond confirmation of CR.

Quality of life is assessed on day 1 of each treatment course (before drug administration) and at 30 days after the completion of study treatment.

Patients are followed at 30 days and then every 3 months for survival.

PROJECTED ACCRUAL: A total of 155 patients (75 for arm I and 80 for arm II) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Locally advanced (stage IIIB) or metastatic (stage IV) disease
  * Inoperable disease
* Relapsed or refractory disease

  * Received 1, and only 1, prior chemotherapy regimen for locally advanced or metastatic disease
* Measurable or evaluable disease
* No symptomatic or inadequately treated brain metastases
* No CNS disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 3 months

Hematopoietic

* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.0 g/dL
* Absolute neutrophil count greater than 1,500/mm^3

Hepatic

* AST and ALT less than 3 times upper limit of normal (ULN)
* Bilirubin less than 1.5 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal

* Creatinine less than 1.8 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* No poorly controlled hypertension

Immunologic

* No active systemic infection requiring treatment
* No prior allergic reaction attributable to compounds containing boron or mannitol
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No peripheral neuropathy grade 2 or greater
* No diabetes mellitus
* No other serious medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 6 weeks since prior monoclonal antibody therapy
* No concurrent routine use of colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy
* No prior docetaxel

  * Prior paclitaxel allowed
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent corticosteroids (e.g., prednisone or prednisolone) except dexamethasone as premedication

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery
* No concurrent surgery for cancer management or treatment

Other

* More than 5 years since prior treatment for any other cancer except basal cell skin cancer or carcinoma in situ of the cervix
* More than 4 weeks since prior investigational agents
* No prior bortezomib
* No other concurrent investigational agents
* No other concurrent clinical research study participation
* No other concurrent antineoplastic therapy
* No concurrent routine use of anti-inflammatory drugs, including cyclo-oxygenase inhibitors (e.g., celecoxib or rofecoxib)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-05; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan H. Schiller, MD, Principal Investigator — University of Wisconsin, Madison
Locations (21):
- United States (21):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Kansas City Cancer Centers - Central, Kansas City, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Fanucchi MP, Fossella FV, Belt R, Natale R, Fidias P, Carbone DP, Govindan R, Raez LE, Robert F, Ribeiro M, Akerley W, Kelly K, Limentani SA, Crawford J, Reimers HJ, Axelrod R, Kashala O, Sheng S, Schiller JH. Randomized phase II study of bortezomib alone and bortezomib in combination with docetaxel in previously treated advanced non-small-cell lung cancer. J Clin Oncol. 2006 Nov 1;24(31):5025-33. doi: 10.1200/JCO.2006.06.1853. PMID 17075122